CLINICAL TRIAL: NCT03096873
Title: Effectiveness of Combined Resistance and Aerobic Exercise Training on Obesity in Adolescent Girls
Brief Title: Combined Resistance and Aerobic Exercise Training on Obesity in Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University (Other)
Collaborators: Dong-Eui University (Other)
Responsible Party: Principal Investigator, Won-mok son, Principal Investigator, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UNOmaha7
Record Dates: First submitted 2017-03-17; First posted 2017-03-30 (Actual); Results first posted 2019-08-19 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Exercise (CON) (No Intervention): Twenty obese adolescent girls. This arm did not perform any exercise training for 12 weeks. Caloric intake: 1921.7 kcal/day
- Exercise (EX) (Experimental): Twenty obese adolescent girls. This arm performed combined exercise training 5 times a week for 12 weeks. Caloric intake: 1921.7 kcal/day
  Interventions: Behavioral: Combined Exercise Training

INTERVENTIONS:
Behavioral: Combined Exercise Training — The combined exercise training were consisted with 5 minutes of warm-up, 20 minutes of resistant band exercises (Upper: seated rows, biceps curl, shoulder flexion, elbow flexion, pushup; Lower: hip flexion, hip extension, calf raise, leg press, squat), 30 minutes of treadmill walking, and 5 minutes of cool-down. Intensity of the training was gradually increased from 40-50% heart rate reserve in 1-4 weeks to 60-70% HRR in 9-12 weeks.
  Arms: Exercise (EX)

SUMMARY:
The purpose of the study was to observe therapeutic effects of combined resistance and aerobic exercise training (CRAE) on hyperinsulemia in obese adolescent girls. Forty obese adolescent girls (14±1 years) participated in this study. The participants were randomly separated into two groups; no-exercise group (n=20) and exercise group (n=20). The exercise group performed 12 weeks of CRAE.

ELIGIBILITY:
Inclusion Criteria:

* Obese with Hyperinsulinemia
* Obese with Abdominal obesity

Exclusion Criteria:

* Hypertension
* Pregnancy
* Chronic diseases
* Weight loss diet within the last 6 months

Ages: 14 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2011-03-03 (Actual); Primary Completion 2011-06-03 (Actual); Study Completion 2011-06-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- No Exercise (CON): Twenty obese adolescent girls. This arm did not perform any exercise training for 12 weeks. Caloric intake: 1921.7 kcal/day (n = 20)
- Exercise (EX): Twenty obese adolescent girls. This arm performed combined exercise training 5 times a week for 12 weeks. Caloric intake: 1921.7 kcal/day (n = 20)
  Combined Exercise Training: The combined exercise training were consisted with 5 minutes of warm-up, 20 minutes of resistant band exercises (Upper: seated rows, biceps curl, shoulder flexion, elbow flexion, pushup; Lower: hip flexion, hip extension, calf raise, leg press, squat), 30 minutes of treadmill walking, and 5 minutes of cool-down. Intensity of the training was gradually increased from 40-50% heart rate reserve in 1-4 weeks to 60-70% HRR in 9-12 weeks.
Period: Overall Study
Arm/Group | No Exercise (CON) | Exercise (EX)
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Exercise (CON) | Exercise (EX) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (1) | 14 (1) | 14 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 20 | 20 | 40
Weight [Mean (Standard Deviation); unit: kilograms] | 75.6 (2.8) | 76.4 (2.8) | 76 (2.8)
Waist circumference [Mean (Standard Deviation); unit: centimeters] | 87.3 (1.5) | 87.6 (0.7) | 87.5 (1.1)
Percentage of body fat [Mean (Standard Deviation); unit: percent] | 43.4 (2.2) | 43 (2.3) | 43.2 (2.2)
Glucose [Mean (Standard Deviation); unit: mmol/L] | 5.6 (0.2) | 5.5 (0.1) | 5.6 (0.2)
Insulin [Mean (Standard Deviation); unit: uU/mL] | 26.2 (3.2) | 27.4 (2.2) | 26.8 (2.7)
Resting heart rate [Mean (Standard Deviation); unit: beats per minute] | 68 (3) | 68 (2) | 68 (3)
Arterial stiffness [Mean (Standard Deviation); unit: m/s] | 8.3 (1) | 8.5 (1.2) | 8.4 (1.1)
Height [Mean (Standard Deviation); unit: meters] | 1.58 (0.13) | 1.6 (0.01) | 1.59 (.07)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30 (1.2) | 30 (2.2) | 30 (1.7)
Blood pressure [Mean (Standard Deviation); unit: mmHg] | 122 (1.2) | 121 (1.4) | 122 (1.3)
Lean body mass [Mean (Standard Deviation); unit: percent] | 43.7 (1.7) | 41.7 (1.4) | 42.7 (1.6)
Leptin [Mean (Standard Deviation); unit: ng/mL] | 21.2 (2.4) | 20.8 (2.1) | 21.0 (2.3)
Adiponectin [Mean (Standard Deviation); unit: ug/mL] | 5.3 (0.8) | 5.7 (0.5) | 5.5 (0.7)
Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) [Mean (Standard Deviation); unit: HOMA-IR Score] — HOMA-IR calculation: fasting insulin (uU/L) x fasting glucose (nmol/L)/22.5 Lower values for this measurement are favorable.
  HOMA-IR Score | 6.4 (0.4) | 6.7 (0.5) | 6.6 (0.5)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 122 (1.3) | 121 (1.4) | 121.2 (1.3)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 80 (2.2) | 80 (1.6) | 80 (1.8)
Volume of maximal oxygen consumption (VO2max) [Mean (Standard Deviation); unit: mL/kg/min of oxygen] — Volume of maximal oxygen consumption (VO2max) was determined using a maximal treadmill test.
  mL/kg/min of oxygen | 25 (2.4) | 25 (1.7) | 25 (2.2)
Arterial stiffness [Mean (Standard Deviation); unit: meters per second (m/s)] — Brachial-ankle Pulse Wave Velocity (m/s) was measured using applanation tonometry.
  meters per second (m/s) | 8.3 (1.4) | 8.5 (1.2) | 8.4 (1.3)
Maximal Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 202 (3) | 203 (4) | 203 (3)

OUTCOME MEASURES:

1. Primary Outcome: Height in Meters
Description: Height was measured before and after 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | No Exercise (CON) | Exercise (EX)
Number analyzed (Participants) | 20 | 20
meters | 1.58 (0.15) | 1.60 (0.11)

2. Primary Outcome: Weight in Kilograms
Description: Weight was measured before and after 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | No Exercise (CON) | Exercise (EX)
Number analyzed (Participants) | 20 | 20
kilograms (kg) | 75.8 (1.5) | 70.2 (2.9)

3. Primary Outcome: BMI in Weight (Kilograms)/Height (Meters)^2
Description: BMI was calculated with weight and height before and after 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kilograms per meter squared (kg/m^2)
Arm/Group | No Exercise (CON) | Exercise (EX)
Number analyzed (Participants) | 20 | 20
kilograms per meter squared (kg/m^2) | 30 (1.4) | 27 (2.1)

4. Primary Outcome: Body Fat in Percents
Description: Body fat was measured before and after 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | No Exercise (CON) | Exercise (EX)
Number analyzed (Participants) | 20 | 20
percent | 43 (2.2) | 39.6 (2.1)

5. Primary Outcome: Lean Body Mass in Percents
Description: Lean body mass was measured before and after 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | No Exercise (CON) | Exercise (EX)
Number analyzed (Participants) | 20 | 20
percent | 43 (2.2) | 39.6 (2.1)

6. Primary Outcome: Waist Circumference in Centimeters
Description: Waist circumference was measured before and after 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | No Exercise (CON) | Exercise (EX)
Number analyzed (Participants) | 20 | 20
centimeters (cm) | 88.2 (1.0) | 83.5 (0.5)

7. Primary Outcome: Glucose Levels in Millimole Per Liter
Description: Glucose levels were measured before and after 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | No Exercise (CON) | Exercise (EX)
Number analyzed (Participants) | 20 | 20
mmol/L | 5.4 (0.1) | 4.3 (0.2)

8. Primary Outcome: Insulin Levels in Micro Unit Per Milliliter
Description: Insulin levels were measured before and after 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: uU/mL
Arm/Group | No Exercise (CON) | Exercise (EX)
Number analyzed (Participants) | 20 | 20
uU/mL | 27 (2.4) | 10.3 (2.1)

9. Primary Outcome: Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: Homeostasis model assessment of Insulin Resistance (HOMA-IR) was calculated before and after 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: HOMA-IR Score
Arm/Group | No Exercise (CON) | Exercise (EX)
Number analyzed (Participants) | 20 | 20
HOMA-IR Score | 6.5 (0.6) | 1.9 (0.7)

10. Primary Outcome: Leptin Levels in Nano Grams Per Milliliter
Description: Leptin levels were measured before and after 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | No Exercise (CON) | Exercise (EX)
Number analyzed (Participants) | 20 | 20
ng/mL | 22.5 (2.3) | 12.8 (1.4)

11. Primary Outcome: Adiponectin Levels in Micro Grams Per Milliliter
Description: Adiponectin levels were measured before and after the training.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | No Exercise (CON) | Exercise (EX)
Number analyzed (Participants) | 20 | 20
ug/mL | 5.7 (0.5) | 8.5 (0.1)

12. Secondary Outcome: Volume of Maximal Oxygen Consumption (VO2max)
Description: Volume of maximal oxygen consumption (VO2max) was determined using a maximal treadmill test before and after 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mL/kg/min of oxygen
Arm/Group | No Exercise (CON) | Exercise (EX)
Number analyzed (Participants) | 20 | 20
mL/kg/min of oxygen | 26 (2.1) | 27 (1.2)

13. Secondary Outcome: Arterial Stiffness
Description: Brachial-ankle Pulse Wave Velocity (m/s) was measured using applanation tonometry before and after 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Arm/Group | No Exercise (CON) | Exercise (EX)
Number analyzed (Participants) | 20 | 20
meters per second (m/s) | 8.4 (1) | 8.4 (1)

14. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure was measured before and after 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | No Exercise (CON) | Exercise (EX)
Number analyzed (Participants) | 20 | 20
mmHg | 124 (1.4) | 120 (0.4)

15. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure was measured before and after 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | No Exercise (CON) | Exercise (EX)
Number analyzed (Participants) | 20 | 20
mmHg | 80 (2.4) | 78 (1.55)

16. Secondary Outcome: Maximal Heart Rate
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | No Exercise (CON) | Exercise (EX)
Number analyzed (Participants) | 20 | 20
beats per minute | 202 (4) | 202 (3)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | No Exercise (CON) | Exercise (EX)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes